CLINICAL TRIAL: NCT02715518
Title: Comparison of Clinical Outcomes Between Fractional Flow Reserve-guided Strategy and Angiography-guided Strategy in Treatment of Non-Infarction Related Artery Stenosis in Patients With Acute Myocardial Infarction
Brief Title: FFR Versus Angiography-Guided Strategy for Management of AMI With Multivessel Disease
Acronym: FRAME-AMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Inje University (Other); Keimyung University Dongsan Medical Center (Other); Sejong General Hospital (Other); Wonju Severance Christian Hospital (Other); Chungbuk National University Hospital (Other); Chosun University Hospital (Other); Inha University Hospital (Other); Gyeongsang National University Hospital (Other); KangWon National University Hospital (Other); Incheon St.Mary's Hospital (Other); Uijeongbu St. Mary Hospital (Other); Ajou University School of Medicine (Other); Chonnam National University Hospital (Other); Kosin University Gospel Hospital (Other); Samsung Changwon Hospital (Other); Kangbuk Samsung Hospital (Other); Yeungnam University Hospital (Other)
Responsible Party: Principal Investigator, Joo-Yong Hahn, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FRAME16453143
Record Dates: First submitted 2016-03-16; First posted 2016-03-22 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute ST-segment elevation myocardial infarction; Acute myocardial infarction; Fractional flow reserve; Percutaneous coronary intervention; Multivessel disease; STEMI; NSTEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Clinical event adjudication and statistical analysis will be blindly performed by independent investigators.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FFR-guided strategy arm (Active Comparator): FFR measurement for non-IRA stenosis (>50% visual estimation) will be performed by continuous infusion of adenosine (140~180ug/kg/min) or intracoronary nicorandil (2mg bolus) injection. The FFR ≤ 0.80 will be targeted for PCI using 2nd generation drug-eluting stent. In case of non-IRA stenosis > 90%, we will judge FFR value of ≤ 0.80.
  The evaluation of non-IRA stenosis by FFR will be recommended to perform during same intervention with primary PCI for IRA. However, exceptions can be made for complex lesions including ACC/AHA classification B2/C lesion where the operator estimates that the revascularization procedure will require significant contrast overload which may lead to deterioration of cardiac and renal function of the patient. Such procedures can be performed in a staged procedure during the same hospitalization.
  Interventions: Device: PCI using 2nd generation drug-eluting stent
- Angiography-guided strategy arm (Active Comparator): Non-IRA stenosis with > 50% stenosis will be the target of PCI using 2nd generation drug-eluting stent.
  As for the angiography-guided strategy arm, PCI for non-IRA stenosis will be recommended during same procedure. However, exceptions can be made for complex lesions including ACC/AHA classification B2/C lesion where the operator estimates that the revascularization procedure will require significant contrast overload which may lead to deterioration of cardiac and renal function of the patient. Such procedures can be performed in a staged procedure during the same hospitalization.
  Interventions: Device: PCI using 2nd generation drug-eluting stent

INTERVENTIONS:
Device: PCI using 2nd generation drug-eluting stent — Percutaneous coronary intervention (PCI) using 2nd generation drug-eluting stent for non-IRA stenosis will be decided according to the allocated arms.
  1. FFR-guided strategy arm
  2. Angiography-guided strategy arm

SUMMARY:
The aim of the study is to compare clinical outcomes following fractional flow reserve (FFR)-guided versus angiography only guided strategy in treatment of non-infarction related artery (non-IRA) stenosis in patients with acute myocardial infarction (AMI) with multivessel disease

Prospective, open-label, randomized, multicenter trial to test the clinical outcomes following FFR-guided or angiography-guided strategy in treatment of non-IRA stenosis in patients with acute AMI with multivessel disease.

DETAILED DESCRIPTION:
The presence of ischemia is a prerequisite for the improvement of clinical outcomes with percutaneous coronary intervention (PCI). It is well-known that the discrepancy exists between angiographic stenosis severity and the presence of myocardial ischemia. This discrepancy cannot completely overcome with even more precise invasive imaging modalities such as intravascular ultrasound or optical coherence tomography.

Currently, fractional flow reserve (FFR) is regarded as a gold-standard invasive method to define lesion-specific ischemia and FFR-guided PCI has been proven to reduce unnecessary revascularization and to enhance patient's clinical outcomes. Therefore, current guidelines recommend FFR measurement for intermediate coronary stenosis when there is no definite evidence of lesion-specific ischemia.

However, previous evidences which well demonstrated the benefit of FFR-guided strategy were mostly generated from non-acute myocardial infarction patients.1, 3-5 Recently FAMOUS-NAMI trial evaluated 176 patients with acute non-ST elevation myocardial infarction (NSTEMI) with multivessel disease, and demonstrated feasibility of FFR measurement in acute NSTEMI patients and also presented that FFR-guided decision making for non-infarct related artery (IRA) stenosis was significantly reduced unnecessary stent implantation without any difference in major adverse cardiovascular events at 1-year as well as medical cost, compared with angiography-only guided decision making process.

Nevertheless, there have been no evidence in clinical setting of acute myocardial infarction (AMI). Since about 30-50% of patients with AMI possess multivessel disease, the ability to accurately assess the functional significance of non-IRA stenoses at the time of initial primary PCI would potentially facilitate revascularization decisions with potential for health and economic benefit. Moreover, avoiding unnecessary stent implantation for non-IRA stenoses in patients with AMI with multivessel disease would reduce the possibility of stent- or procedure related complications, and enhance long-term prognosis of patients.

Therefore, the FRAME-AMI trial will compare clinical outcomes after index primary PCI between FFR-guided strategy versus angiography only-guided strategy for management of non-IRA stenoses in AMI with multivessel disease patients.

ELIGIBILITY:
(1) Inclusion Criteria

1. Subject must be at least 19 years of age
2. Acute ST-segment elevation myocardial infarction (STEMI) A. ※ STEMI: "ST-segment elevation ≥0.1 mV in ≥2 contiguous leads B. or documented newly developed left bundle-branch block "
3. Acute non-ST-segment elevation myocardial infarction (NSTEMI)

   A. ※ NSTEMI: NSTEMI is defined as a combination of criteria with mandated elevation of a cardiac biomarker, preferably high-sensitive cardiac troponin with at least one value above 99th percentile of the upper reference limit and at least one of the following:
4. Symptoms of ischaemia.
5. New or presumed new significant ST-T wave changes
6. Development of pathological Q waves on electrocardiography (ECG).
7. Imaging evidence of new or presumed new loss of viable myocardium or regional wall motion abnormality.
8. Intracoronary thrombus detected on angiography.
9. Primary percutaneous coronary intervention (PCI) in < 12 h after the onset of symptoms for STEMI patients (In case of NSTEMI, PCI should be performed within 72 hours of symptom onset)
10. Multivessel disease (at least one stenosis of >50% in a non-culprit vessel ≥ 2.0 mm by visual estimation)
11. Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving invasive physiologic evaluation and PCI and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.

(2) Exclusion criteria

1. Severe stenosis with TIMI flow ≤ II of the non-IRA artery
2. Unprotected left main coronary artery disease (stenosis > 50% by visual estimation)
3. Non-IRA stenosis not amenable for PCI treatment by operators' decision)
4. Chronic total occlusion in non-IRA
5. Cardiogenic shock (Killip class IV) already at presentation or the completion of IRA PCI
6. Intolerance to Aspirin, Clopidogrel, Plasugrel, Ticagrelor, Heparin, Bivaluridin, or Everolimus, Zotarolimus
7. Known true anaphylaxis to contrast medium (not allergic reaction but anaphylactic shock)
8. Pregnancy or breast feeding
9. Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
10. Other primary valvular disease with severe degree: severe mitral regurgitation, mitral stenosis, severe aortic regurgitation, or aortic stenosis
11. Patients with a history of Coronary Artery Bypass Graft (CABG) or treated with fibrinolytic Therapy
12. Unwillingness or inability to comply with the procedures described in this protocol.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1292 (Actual)
Dates: Start 2016-08-19 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Patient-oriented composite outcome | 24 months
  a composite of death, myocardial infarction, or repeat revascularization

SECONDARY OUTCOMES:
All-cause mortality | 24 months
  All-cause mortality
Cardiac death | 24 months
  Cardiac death
Any myocardial infarction without procedure-related myocardial infarction | 24 months
  Any myocardial infarction without procedure-related myocardial infarction
Any myocardial infarction with periprocedural myocardial infarction | 24 months
  Any myocardial infarction with periprocedural myocardial infarction
Any revascularization | 24 months
  ischemia-driven or all
Infarct-related artery (IRA) repeat revascularization | 24 months
  ischemia-driven or all
Non-IRA repeat revascularization | 24 months
  ischemia-driven or all
Stent thrombosis | 24 months
  ARC-defined definite stent thrombosis
Stroke | 24 months
  ischemic and hemorrhagic
Total amount of contrast use | 1 week
  From primary PCI to end of the procedure including amount of staged procedure
Incidence of contrast-induced nephropathy | 3 days
  defined as an increase in serum creatinine of ≥0.5mg/dL or ≥25% from baseline within 48-72 hours after contrast agent exposure
Seattle Angina Questionnaires | 12-month
  Angina severity
Seattle Angina Questionnaires | 24-month
  Angina severity
All-cause death and myocardial infarction | 24-month
  A composite of all-cause death and any myocardial infarction (MI) according to the ARC consensus
Death, spontaneous myocardial infarction, or repeat revascularization | 24-month
  A composite of Death, spontaneous myocardial infarction, or repeat revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Yong Hahn, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked
Supporting Information: Study Protocol, SAP
Time Frame: After reporting of the main results.
Access Criteria: After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked

REFERENCES:
- [Derived] Lee SH, Kim H, Lee JM, Ahn JH, Park S, Lee YK, Joo D, Cho KH, Kim MC, Sim DS, Kim HK, Park KH, Choo EH, Kim CJ, Ahn SG, Doh JH, Lee SY, Park SD, Lee HJ, Kang MG, Nam CW, Hong D, Joh HS, Choi KH, Park TK, Yang JH, Song YB, Choi SH, Kim JH, Ahn Y, Jeong MH, Gwon HC, Hahn JY, Koh JS, Hong YJ; FRAME-AMI Investigators. Clinical Relevance of Fractional Flow Reserve-Guided Percutaneous Coronary Interevention According to Left Ventricular Ejection Fraction in Patients With Acute Myocardial Infarction and Multivessel Disease. J Am Heart Assoc. 2025 Sep 2;14(17):e043414. doi: 10.1161/JAHA.125.043414. Epub 2025 Aug 29. PMID 40878980
- [Derived] Lim Y, Jang J, Lee SH, Ahn JH, Hong YJ, Ahn Y, Jeong MH, Kim CJ, Hahn JY, Lee JM, Park KH, Choo EH, Ahn SG, Doh JH, Lee SY, Park SD, Lee HJ, Kang MG, Cho YK, Nam CW, Bu SH, Kim MC. Staged versus immediate complete revascularization for non-culprit arteries in acute myocardial infarction: a post-hoc analysis of FRAME-AMI. Front Cardiovasc Med. 2024 Dec 12;11:1475483. doi: 10.3389/fcvm.2024.1475483. eCollection 2024. PMID 39726942
- [Derived] Kwon W, Choi KH, Lee SH, Hong D, Shin D, Kim HK, Park KH, Choo EH, Kim CJ, Kim MC, Hong YJ, Ahn SG, Doh JH, Lee SY, Park SD, Lee HJ, Kang MG, Koh JS, Cho YK, Nam CW, Joh HS, Kyu Park T, Yang JH, Song YB, Choi SH, Jeong MH, Gwon HC, Hahn JY, Lee JM; FRAME-AMI Investigators. Clinical Value of Single-Projection Angiography-Derived FFR in Noninfarct-Related Artery. Circ Cardiovasc Interv. 2024 May;17(5):e013844. doi: 10.1161/CIRCINTERVENTIONS.123.013844. Epub 2024 May 21. PMID 38771911
- [Derived] Hong D, Lee SH, Lee J, Lee H, Shin D, Kim HK, Park KH, Choo EH, Kim CJ, Kim MC, Hong YJ, Jeong MH, Ahn SG, Doh JH, Lee SY, Don Park S, Lee HJ, Kang MG, Koh JS, Cho YK, Nam CW, Choi KH, Park TK, Yang JH, Song YB, Choi SH, Gwon HC, Guallar E, Cho J, Hahn JY, Kang D, Lee JM; FRAME-AMI Investigators. Cost-Effectiveness of Fractional Flow Reserve-Guided Treatment for Acute Myocardial Infarction and Multivessel Disease: A Prespecified Analysis of the FRAME-AMI Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2352427. doi: 10.1001/jamanetworkopen.2023.52427. PMID 38270954
- [Derived] Seung J, Choo EH, Kim CJ, Kim HK, Park KH, Lee SH, Kim MC, Hong YJ, Ahn SG, Doh JH, Lee SY, Park SD, Lee HJ, Kang MG, Koh JS, Cho YK, Nam CW, Koo BK, Lee BK, Yun KH, Hong D, Joh HS, Choi KH, Park TK, Lee JM, Yang JH, Song YB, Choi SH, Gwon HC, Hahn JY; FRAME-AMI Investigators. Angiographic Severity of the Nonculprit Lesion and the Efficacy of Fractional Flow Reserve-Guided Complete Revascularization in Patients With AMI: FRAME-AMI Substudy. Circ Cardiovasc Interv. 2024 Jan;17(1):e013611. doi: 10.1161/CIRCINTERVENTIONS.123.013611. Epub 2023 Nov 6. PMID 37929584
- [Derived] Lee SH, Hong D, Shin D, Kim HK, Park KH, Choo EH, Kim CJ, Kim MC, Hong YJ, Ahn SG, Doh JH, Lee SY, Park SD, Lee HJ, Kang MG, Koh JS, Cho YK, Nam CW, Joh HS, Choi KH, Park TK, Yang JH, Song YB, Choi SH, Jeong MH, Gwon HC, Hahn JY, Lee JM; FRAME-AMI Investigators. QFR Assessment and Prognosis After Nonculprit PCI in Patients With Acute Myocardial Infarction. JACC Cardiovasc Interv. 2023 Oct 9;16(19):2365-2379. doi: 10.1016/j.jcin.2023.08.032. PMID 37821181
- [Derived] Lee JM, Kim HK, Park KH, Choo EH, Kim CJ, Lee SH, Kim MC, Hong YJ, Ahn SG, Doh JH, Lee SY, Park SD, Lee HJ, Kang MG, Koh JS, Cho YK, Nam CW, Koo BK, Lee BK, Yun KH, Hong D, Joh HS, Choi KH, Park TK, Yang JH, Song YB, Choi SH, Gwon HC, Hahn JY; FRAME-AMI Investigators. Fractional flow reserve versus angiography-guided strategy in acute myocardial infarction with multivessel disease: a randomized trial. Eur Heart J. 2023 Feb 7;44(6):473-484. doi: 10.1093/eurheartj/ehac763. PMID 36540034
- [Derived] Shin D, Rhee TM, Lee SH, Lee JM. Revascularization Strategies in Patients With ST-Segment Elevation Myocardial Infarction and Multivessel Disease: Is FFR-Guided Strategy Still Valuable? Korean Circ J. 2022 Apr;52(4):280-287. doi: 10.4070/kcj.2021.0416. PMID 35388996